CLINICAL TRIAL: NCT03862547
Title: Role and Clinical Relevance of Nerve Growth Factor (NGF) and Its Receptors (TrKA and p75NTR) in Patients With Erectile Dysfunction and Diabetes With or Wothout Metabolic Syndrome
Brief Title: NGF, TrKA,p75NTR in Men With ED and Diabetes With or Without MS
Acronym: ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Collaborators: Ester Illiano, MD (Unknown); Mario Rende,Full Professor (Unknown); Alessandra Psitilli, Researcher (Unknown); Anna Stabile, Researcher (Unknown)
Responsible Party: Principal Investigator, Elisabetta Costantini, Associate Professor,MD, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DE1
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; NGF; TrKA; p75NTR
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with ED and diabetes (Experimental): A peripheral blood sample from the cubital vein
  1. A collection of peripheral blood from the routinary cubital vein for hormone dosage and metabolic evaluation
  2. An introverted cavernous infiltration of Prostaglandin E1 to achieve erection (Aprostadil);
  3. A blood sample from both the corpus cavernosum and the cubital vein, once the erection is achieved Baseline interaction of prostaglandin E1 on the concentration of NGF released in the medium and on the expression of its receptors Evaluation of NGF and Cytokine levels Expression analysis of TrKA and p75NTR receptors and intracellular cytokines in PBMCs
  Interventions: Diagnostic Test: A peripheral blood sample from the cubital vein

INTERVENTIONS:
Diagnostic Test: A peripheral blood sample from the cubital vein — Evaluation of NGF and Cytokine levels A portion of each blood sample and medium conditioned by PBMC will be used for the enzyme immunoassay of NGF and pro and anti-inflammatory cytokine levels (TNF alfa and IL-10).
  Expression analysis of TrKA and p75NTR receptors and intracellular cytokines in PBMCs The remaining part of each blood sample and PBMC of the in vitro experiment will be used for the cytofluorimetric evaluation of the expression of TrKA, p75NTR and the pro and anti-inflammatory cytokines and reactive oxygen species.
  Other Names: cavernous infiltration of PGE1

SUMMARY:
To evaluate the level of NGF,TrKA and p75NTR in patientd with erectile dysfunction and diabetes with or without metabolic syndrome

DETAILED DESCRIPTION:
Penile erection is a complex phenomenon which implies a delicate and co-ordinated equilibrium among the neurological, vascular and the smooth muscle compartment. It includes arterial dilation, trabecular smooth muscle relaxation and activation of the corporeal veno-occlusive mechanism. Erectile Dysfunction (ED) is defined as the persistent inability to attain and maintain an erection sufficient to permit satisfactory sexual performance. Erectile Dysfunction may affect physical and psychosocial health and may have a significant impact on the quality of life (QoL) of sufferers and their partner's . There is increasing evidence that ED can be an early manifestation of coronary artery and peripheral vascular disease. Erectile Dysfunction should not be regarded only as a QoL issue, but also as a potential warning sign of cardiovascular disease (CVD) .The most important organic causes of ED are vascular, metabolic, neurogenic, hormonal and pharmacological. 35-90% of diabetic patients suffer from ED In the latter metabolic disease, Dai et al. have identified as a possible etiology of ED a lack of interaction between nerve growth factor (NGF) and its TrKA receptor, resulting in a noticeable increase in NGF levels in the corpora cavernosa11. Furthermore, Hou et al. have shown that the activation of the NGF / TrKA system in the corpora cavernosa (increased expression of NGF and TrKA mRNA and upregulation of c-raf, ERK1 / 2 and CREB1) improves erectile function in mice with ED and diabetes mellitus.

The objectives of this study are:

* The primary outcome is to evaluate the systemic plasma concentration and the concentration in cavernous bodies of penis of NGF in patients with ED and diabetes with or without metabolic syndrome (a); (b) the expression of its TrKA and p75NTR receptors in the mononuclear cells taken from peripheral blood and in cavernous bodies of penis.
* The secondary outcome is to evaluate whether the levels of NGF and its receptors in the mononuclear cells can correlate with the clinical staging of ED.

Prospective pilot study. 12 patients diagnosed with ED with diabetes with or without metabolic syndrome( Mets )aged between 18 and 65 will be recruited. Each patient will undergo an initial evaluation that includes: the pathological and pharmacological anamnesis, the local objective examination and the compilation of the validated questionnaire International Index of Erectile Function Questionnaire short form (IIEF5).

Based on the IIEF5 score, patients will be divided into 4 groups (each of 10 patients):

1. mild ED (score 17-21)
2. mild to moderate ED (score 12-16)
3. Moderate ED (score 8-11)
4. Severe ED (score 5-7)

In vivo study:

Each patient will then be submitted in succession to:

1. A collection of peripheral blood from the routinary cubital vein for hormone dosage Follicle-stimulating hormone (FSH), Luteinizing hormone (LH), TESTOSTERONE FREE AND TOTAL, ESTRADIOL, PROLACTIN) and metabolic evaluation (total HDL cholesterol, LDH, glycemia, lipidemic framework); and an aliquot will be used for in vitro study
2. An introverted cavernous infiltration of Prostaglandin E1 to achieve erection (Aprostadil);
3. A blood sample from both the corpus cavernosum and the cubital vein, once the erection is achieved

Vitro study To verify a possible baseline interaction of prostaglandin E1 on the concentration of NGF released in the medium and on the expression of its receptors, an in vitro study will be performed using mononuclear cells isolated from peripheral blood (PBMC) obtained from buffy coat treated with prostaglandin E1

Evaluation of NGF and Cytokine levels A portion of each blood sample and medium conditioned by PBMC will be used for the enzyme immunoassay of NGF and pro and anti-inflammatory cytokine levels (TNF alfa and IL-10).

Expression analysis of TrKA and p75NTR receptors and intracellular cytokines in PBMCs.

The remaining part of each blood sample and PBMC of the in vitro experiment will be used for the cytofluorimetric evaluation of the expression of TrKA, p75NTR and the pro and anti-inflammatory cytokines and reactive oxygen species

Evaluation of the levels of NGF and its receptors in the different degrees of severity of the EDThe levels of NGF and its receptors will be stratified into the 4 groups of clinical severity of the ED

In vitro study An in vitro study will be performed using PBMC obtained from buffy coat of healthy subjects treated with prostaglandin E1.

Statistical analysis of the results The data obtained during the study will be treated with appropriate statistical tests. The results will be expressed in terms of mean ± standard error and compared by appropriate statistical tests (ANOVA or non-parametric where appropriate).

Expected results From the present study we expect to obtain more information on the impact and relevance of the NGF / TrKA / p75NTR pathway on DE in patients with Mets. Furthermore, we expect a correlation between the plasma levels of NGF and its receptors in relation to the clinical severity of the ED.

ELIGIBILITY:
Inclusion Criteria:

* men with DE and metabolic syndrome

Exclusion Criteria:

* men with DE without metabolic syndrome

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men with erectile dysfunction and metabolic syndrome
Enrollment: 40 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Baseline NGF | baseline
  plasmatic concentration
intracavernous NGF | 15 minutes
  intracavernous concetration
plasmatic NGF | 15 minutes
  plasmatic concetration
Baseline TRka | baseline
  plasmatic concetration
plasmatic TRka | 15 minutes
  plasmatic concetration
Intracavernous TRka | 15 minutes
  intracavernous concetration
Baseline p75NTR | baseline
  plasmatic concentration
plasmatic p75NTR | 15 minutes
  plasmatic concentration
intracavernous p75NTR | 15 minutes
  intracavernous concentration

SECONDARY OUTCOMES:
plasmatic concentration verus intracavernous concetration | 15 minutes
  to evaluate any differences between the data obtained from the systemic levy versus the intracavernous sampling.
clinical staging of ED and NGF,TrKa,p75NTR | 15 minutes
  is to evaluate if the levels of NGF and its receptors in the mononuclear cells can correlate with the clinical staging of ED.

CONTACTS AND LOCATIONS:
Overall Officials: Ester Illiano, MD, Study Director — University Of Perugia
Locations (1):
- Elisabetta Costantini, Terni, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teng KK, Hempstead BL. Neurotrophins and their receptors: signaling trios in complex biological systems. Cell Mol Life Sci. 2004 Jan;61(1):35-48. doi: 10.1007/s00018-003-3099-3. PMID 14704852
- [Background] Arcidiacono P, Stabile AM, Ragonese F, Pistilli A, Calvieri S, Bottoni U, Crisanti A, Spaccapelo R, Rende M. Anticarcinogenic activities of sulforaphane are influenced by Nerve Growth Factor in human melanoma A375 cells. Food Chem Toxicol. 2018 Mar;113:154-161. doi: 10.1016/j.fct.2018.01.051. Epub 2018 Jan 31. PMID 29407470
- [Background] Pistilli A, Rende M, Crispoltoni L, Montagnoli C, Stabile AM. LY294002 induces in vitro apoptosis and overexpression of p75NTR in human uterine leiomyosarcoma HTB 114 cells. Growth Factors. 2015;33(5-6):376-83. doi: 10.3109/08977194.2015.1118096. Epub 2015 Dec 10. PMID 26653825
- [Background] Pula G, Pistilli A, Montagnoli C, Stabile AM, Rambotti MG, Rende M. The tricyclic antidepressant amitriptyline is cytotoxic to HTB114 human leiomyosarcoma and induces p75(NTR)-dependent apoptosis. Anticancer Drugs. 2013 Oct;24(9):899-910. doi: 10.1097/CAD.0b013e328364312f. PMID 23872911
- [Background] Rende M, Pistilli A, Stabile AM, Terenzi A, Cattaneo A, Ugolini G, Sanna P. Role of nerve growth factor and its receptors in non-nervous cancer growth: efficacy of a tyrosine kinase inhibitor (AG879) and neutralizing antibodies antityrosine kinase receptor A and antinerve growth factor: an in-vitro and in-vivo study. Anticancer Drugs. 2006 Sep;17(8):929-41. doi: 10.1097/01.cad.0000224459.13651.fd. PMID 16940803
- [Background] Rask-Madsen C, King GL. Mechanisms of Disease: endothelial dysfunction in insulin resistance and diabetes. Nat Clin Pract Endocrinol Metab. 2007 Jan;3(1):46-56. doi: 10.1038/ncpendmet0366. PMID 17179929
- [Background] Jackson G. The importance of risk factor reduction in erectile dysfunction. Curr Urol Rep. 2007 Nov;8(6):463-6. doi: 10.1007/s11934-007-0049-x. PMID 18042325
- [Background] Kaya E, Sikka SC, Gur S. A comprehensive review of metabolic syndrome affecting erectile dysfunction. J Sex Med. 2015 Apr;12(4):856-75. doi: 10.1111/jsm.12828. Epub 2015 Feb 11. PMID 25675988
- [Background] Dai YT, Chen Y, Yao LS, Yang R, Sun ZY, Wen DG. [Expression of nerve growth factor in cavernous tissue and its effects on the treatment of rats with diabetic erectile dysfunction]. Zhonghua Nan Ke Xue. 2005 Oct;11(10):748-51, 754. Chinese. PMID 16281507